CLINICAL TRIAL: NCT04954742
Title: An Open-label, Prospective, Single Centre Study of the Effects of Riociguat on RIght VEntricular Size and Function in Pulmonary Arterial Hypertension and Chronic Thromboembolic Pulmonary Hypertension
Brief Title: Effects of Riociguat on RIght VEntricular Size and Function in PAH and CTEPH
Acronym: RIVERII
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Strategic re-prioritization by the IMP supplier. Decision not safety-related
Sponsor: Heidelberg University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Prof. Dr. med. Ekkehard Gruenig, Head of centre for pulmonary hypertension, Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-06RCT
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Primary Pulmonary Arterial Hypertension; Chronic Thromboembolic Pulmonary Hypertension
Keywords: pulmonary arterial hypertension; Chronic Thromboembolic Pulmonary Hypertension; riociguat; right heart function
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Riociguat (Other): Riociguat (1 mg, 1.5 mg, 2 mg and 2.5 mg three times daily) starting at 1.0 mg three times daily at the beginning of the study. Dosage will be individually up-titrated up to a maximum dosage of 2.5 mg three times daily after 8 weeks. Study medication will be provided orally with or without food. Tablets should be taken three times daily approximately 6 to 8 hours apart.
  Interventions: Drug: Riociguat

INTERVENTIONS:
Drug: Riociguat — Treatment will be initiated and individually adjusted according to systolic blood pressure and tolerability. During the titration phase, each patient will be asked to measure their peripheral systolic blood pressure and the heart rate at home three times per day and document the values in the patient diary. The results will be examined by the investigator during each visit/phone call-visit. Provided that the systolic blood pressure is ≥ 95 mmHg measured at trough before intake of each dose and the patient has no signs or symptoms of hypotension, the dose of study medication will be titrated by +0.5 mg tid every 2 weeks until maximal tolerated dosage (maximal permitted dose: of 2.5 mg tid). After the titration period, blood pressure should be measured upon signs or symptoms of hypotension. Maintenance dose: The established individual dose should be maintained unless signs and symptoms of hypotension occur.
  Other Names: MK-4836; ATC code: C02KX05

SUMMARY:
This is an open-label, single-armed, prospective single-centre clinical study to evaluate the effect of riociguat on right heart size and function in patients with manifest PAH and CTEPH.

DETAILED DESCRIPTION:
Right heart size and function are of utmost prognostic importance in PAH/CTEPH. RV performance measured by echocardiography and enlarged RA area have been shown to be independent prognostic factors in PAH. Recently, a retrospective single centre study has shown that riociguat treatment was associated with a significant reduction of RV and RA area after 3, 6 and 12 months compared to baseline. RA area significantly decreased after 12 months and RV systolic function assessed with tricuspid annular plane systolic excursion (TAPSE) improved after 6 and 12 months of riociguat therapy. The results were confirmed by a recent retrospective multicentre study. It is therefore reasonable to assume a beneficial effect of riociguat on right heart size and function.

The primary efficacy endpoint in this study is the change in RV and RA area from baseline to 24 weeks. Treatment will be initiated and individually adjusted according to systolic blood pressure and tolerability. Patients who discontinue medication prematurely will be asked to continue with study assessments and perform study visits as outlined in the protocol.

Medical examinations comprise medical history, physical examination, electrocardiogram (ECG), blood gas analyses, lung function tests, laboratory testing (including NT-proBNP), echocardiography at rest, and right heart catheterization (RHC) according to clinical practice of the PH centre.

The prospective period of data collection comprises a 24-week study period a follow-up phase of about 30±7 days.

Outcome (survival and transplant-free survival) of all patients will be assessed when the last patient has terminated his/her 24-week observation period.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age at time of inclusion.
2. Male and female patients with symptomatic PAH with a mean pulmonary artery pressure (mPAP) >20 mmHg and pulmonary vascular resistance (PVR) ≥2 Wood Units (WU), pulmonary arterial wedge pressure (PAWP) ≤15 mmHg (Group I / Nice Clinical Classification of Pulmonary Hypertension) or CTEPH (Group IV / Nice Clinical Classification of Pulmonary Hypertension) defined as inoperable measured at least 3 months after start of full anticoagulation and mPAP >20 mmHg and PVR ≥2 WU, PAWP ≤15 mmHg; or with persisting or recurrent PH after pulmonary endarterectomy (mPAP >20 mmHg and PVR ≥2 WU, PAWP ≤15 mmHg measured at least 6 months after surgery (acc. to Simonneau et al. 2018).
3. Treatment naïve patients (with respect to PAH specific medication) and patients pre-treated with an endothelin receptor antagonist or a prostacyclin analogue, pre-treated for 2 months before screening at most (according to upfront combination treatment).*
4. *Pre-treated patients need to be stable on endothelin receptor antagonists or prostacyclin treatment for at least two weeks prior to Visit 1. "Stable" is defined as no change in the type of endothelin receptor antagonists or prostacyclin analogue and the respective daily dose.
5. A patient may also be enrolled, if a persisting phosphodiesterase type 5 (PDE-5) inhibitor treatment (pre-treated for 2 months before screening at most) with or without combination treatment with an endothelin receptor antagonist or prostacyclin analogue is to be switched to riociguat by clinical indication, particularly when the patient´s risk-profile remained in intermediate risk group despite adequate initial treatment including PDE5i (defined as at least 3 of the following parameters: clinical signs of progression, persistent WHO-FC III, 6MWD between 165-440m, peak V02 11-15ml/min/kg (35-65% predicted), NTproBNP 300-1400 ng/l, RA-area 18-26cm2,RAP 8-14mmHg, CI 2,0-2,4 l/min) or in case of PDE5i intolerance. Any decision to switch will be made by the clinicians at a regular clinical follow-up visit.
6. Unspecific treatments which may also be used for the treatment of PH such as oral anticoagulants, diuretics, digitalis, calcium channel blockers or oxygen supplementation are permitted. However, treatment with anticoagulants (if indicated) must have been started at least 1 month before visit in patients with PAH 1.
7. RHC results must not be older than 6 months at screening (will be considered as baseline values) and must have been measured in the participating centre under standardized conditions (refer to the study specific Swan Ganz catheterization manual). If the respective measurements have not been performed in context with the patient's regular diagnostic workup, they have to be performed as a part of the study during the pre-study phase (after the patient signed the informed consent).
8. Women without childbearing potential defined as postmenopausal women aged 50 years or older, women with bilateral tubal ligation, women with bilateral ovariectomy, and women with hysterectomy can be included in the study.
9. Women of childbearing potential can only be included in the study if all of the following applies (listed below): a. Negative serum pregnancy test at Screening and a negative urine pregnancy test at study start (visit 1). b. Agreement to undertake monthly urine pregnancy tests during the study and up to at least 30 days after study treatment discontinuation. These tests should be performed by the patient at home. c. Agreement to follow the contraception scheme as specified from Screening until at least 30 days after study treatment discontinuation.
10. Patients who are able to understand and follow instructions and who are able to participate in the study for the entire period.
11. Patients must have given their written informed consent to participate in the study after having received adequate previous information and prior to any study-specific procedures.

Exclusion Criteria:

1. Pregnant women, or breast-feeding women, or women of childbearing potential not able or willing to comply with study-mandated contraception methods specified above.
2. Patients with PH specific treatment <2 months before screening.
3. Patients with a medical disorder, condition, or history of such that would impair the patient's ability to participate or complete this study in the opinion of the investigator.
4. Patients with underlying medical disorders with an anticipated life expectancy below 2 years (e.g. active cancer disease with localized and/or metastasized tumour mass).
5. Patients with a history of severe or multiple drug allergies
6. Patients with hypersensitivity to the investigational drug or any of the excipients.
7. Patients unable to perform a valid 6MWD test (e.g. orthopaedic disease, peripheral artery occlusive disease, which affects the patient´s ability to walk).
8. The following specific medications for concomitant treatment of PH or medications which may exert a pharmacodynamic interaction with the study drug are not allowed:

   1. Parenteral prostacyclin analogues
   2. Specific phosphodiesterase inhibitors (e.g. sildenafil or tadalafil): may be switched to riociguat but not be given in addition to the study drug
   3. or unspecific phosphodiesterase inhibitors (e.g. dipyridamole, theophylline)
   4. NO donors (e.g. Nitrates)
9. Pulmonary diseases exclusions

   1. Moderate to severe bronchial asthma or COPD (Forced Expiratory Volume <60% predicted) or severe restrictive lung disease (Total Lung Capacity < 70% predicted) and/or defined as if high resolution computed tomography shows <20% parenchymal lung disease.
   2. Severe congenital abnormalities of the lungs, thorax, and diaphragm.
   3. Clinical or radiological evidence of Pulmonary-Veno-Occlusive Disease (PVOD) or Pulmonary Capillary Haemangiomatosis (PCH) or PH and idiopathic interstitial pneumonia (PH-IIP)
10. Cardiovascular exclusions:

    1. Uncontrolled arterial hypertension (systolic blood pressure >180 mmHg and /or diastolic blood pressure >110 mmHg).
    2. Systolic blood pressure <95 mmHg.
    3. Left heart failure with an ejection fraction less than 40%.
    4. Pulmonary venous hypertension with pulmonary arterial wedge pressure >15 mmHg.
    5. Hypertrophic obstructive cardiomyopathy.
    6. Severe proven or suspected coronary artery disease according to investigators opinion (patients with Canadian Cardiovascular Society Angina Classification class 2-4, and/or requiring nitrates, and/or myocardial infarction within the last 3 months before Visit 1).
    7. Clinical evidence of symptomatic atherosclerotic disease (e.g. peripheral artery disease with reduced walking distance, history of stroke with persistent neurological deficit etc).
11. Exclusions related to disorders in organ function:

    a) Clinically relevant hepatic dysfunction indicated by: i. bilirubin >2 times upper limit normal ii. and / or hepatic transaminases >3 times upper limit normal iii. and / or signs of severe hepatic insufficiency (e.g. impaired albumin synthesis with an albumin < 32 g/l, hepatic encephalopathy > grade 1a: West Haven Criteria of Altered Mental Status In Hepatic Encephalopathy) b) Renal insufficiency (glomerular filtration rate <30 ml/min e.g. calculated based on the Cockcroft formula).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Change in RV (right ventricular) area | Baseline to 24 weeks
  echocardiographic analysis right atrial (RA) area, measured by echocardiography.
Change in RA (right atrial) area | Baseline to 24 weeks
  echocardiographic analysis

SECONDARY OUTCOMES:
Change in RV Area | baseline to 12 weeks
  echocardiographic analysis
Change in RA Area | baseline to 12 weeks
  echocardiographic analysis
Change in systolic pulmonary artery pressure (sPAP) | baseline to 12 weeks
  echocardiographic analysis
Change in systolic pulmonary artery pressure (sPAP) | baseline to 24 weeks
  echocardiographic analysis
Change in RV fractional area change (FAC) | baseline to 24 weeks
  echocardiographic analysis
Change in RV fractional area change (FAC) | baseline to 12 weeks
  echocardiographic analysis
Change in Peak velocity of tricuspid regurgitation (TRV) | baseline to 12 weeks
  echocardiographic analysis
Change in Peak velocity of tricuspid regurgitation (TRV) | baseline to 24 weeks
  echocardiographic analysis
Change in inferior vena cava (IVC) diameter and IVC collapse | baseline to 24 weeks
  echocardiographic analysis
Change in inferior vena cava (IVC) diameter and IVC collapse | baseline to 12 weeks
  echocardiographic analysis
Change in Right Ventricle Outflow Tract Velocity Time Integral (RVOT VTI) | baseline to 12 weeks
  echocardiographic analysis
Change in Right Ventricle Outflow Tract Velocity Time Integral (RVOT VTI) | baseline to 24 weeks
  echocardiographic analysis
Change in Eccentricity index (EI) | baseline to 24 weeks
  echocardiographic analysis
Change in Eccentricity index (EI) | baseline to 12 weeks
  echocardiographic analysis
Change in Tricuspid Annular Plane Systolic Excursion (TAPSE) | baseline to 12 weeks
  echocardiographic analysis
Change in Tricuspid Annular Plane Systolic Excursion (TAPSE) | baseline to 24 weeks
  echocardiographic analysis
Change in Right ventricular pump function (qualitative) | baseline to 24 weeks
  echocardiographic analysis
Change in left ventricular pump function (qualitative) | baseline to 24 weeks
  echocardiographic analysis
Change in Right ventricular pump function (qualitative) | baseline to 12 weeks
  echocardiographic analysis
Change in left ventricular pump function (qualitative) | baseline to 12 weeks
  echocardiographic analysis
Change in Left Atrial (LA) diameter | baseline to 12 weeks
  echocardiographic analysis
Change in Left Atrial (LA) diameter | baseline to 24 weeks
  echocardiographic analysis
Change in LV diastolic function | baseline to 24 weeks
  echocardiographic Analysis measured as: (LV transmitral E wave and A wave, E' wave of interventricular septum and lateral wall pulsed tissue Doppler, isovolumic relaxation time, mitral deceleration time)
Change in LV diastolic function | baseline to 12 weeks
  echocardiographic Analysis measured as: (LV transmitral E wave and A wave, E' wave of interventricular septum and lateral wall pulsed tissue Doppler, isovolumic relaxation time, mitral deceleration time)
Change in Diameters of pulmonary artery | baseline to 12 weeks
  echocardiographic Analysis
Change in Diameters of pulmonary artery | baseline to 24 weeks
  echocardiographic Analysis
Change in cardiac index | baseline and after 24 weeks
  Pulmonary hemodynamics by right heart catheterization
Change in cardiac output | baseline and after 24 weeks
  Pulmonary hemodynamics by right heart catheterization
Change in sPAP | baseline and after 24 weeks
  Pulmonary hemodynamics by right heart catheterization
Change in dPAP | baseline and after 24 weeks
  Pulmonary hemodynamics by right heart catheterization
Change in mPAP | baseline and after 24 weeks
  Pulmonary hemodynamics by right heart catheterization
Change in PAWP | baseline and after 24 weeks
  Pulmonary hemodynamics by right heart catheterization
Change in right atrial pressure (RAP) | baseline and after 24 weeks
  Pulmonary hemodynamics by right heart catheterization
Change in PVR | baseline and after 24 weeks
  Pulmonary hemodynamics by right heart catheterization
Change in Central venous saturation from pulmonary artery | baseline and after 24 weeks
  Pulmonary hemodynamics by right heart catheterization
Change in 6-minute walking distance | baseline to 12 weeks
  Change in exercise capacity
Change in 6-minute walking distance | baseline to 24 weeks
  Change in exercise capacity
forced vital capacity (FVC) | baseline to 12 weeks
  Change in Lung function Tests
forced vital capacity (FVC) | baseline to 24 weeks
  Change in Lung function Tests
Change in forced expiratory volume in one second (FEV1) | baseline to 12 weeks
  Change in Lung function Tests
Change in forced expiratory volume in one second (FEV1) | baseline to 24 weeks
  Change in Lung function Tests
Change in FEV1% of maximal vital capacity (VC max) | baseline to 12 weeks
  Change in Lung function Tests
Change in FEV1% of maximal vital capacity (VC max) | baseline to 24 weeks
  Change in Lung function Tests
Change in total lung capacity (TLC) | baseline to 12 weeks
  Change in Lung function Tests
Change in total lung capacity (TLC) | baseline to 24 weeks
  Change in Lung function Tests
Change in residual volume | baseline to 12 weeks
  Change in Lung function Tests
Change in residual volume | baseline to 24 weeks
  Change in Lung function Tests
Change in diffusion-limited carbon monoxide (DLCO) | baseline to 24 weeks
  Change in Lung function Tests
Change in diffusion-limited carbon monoxide (DLCO) | baseline to 12 weeks
  Change in Lung function Tests
Change in DLCO/VA (Krogh) factor | baseline to 12 weeks
  Change in Lung function Tests
Change in DLCO/VA (Krogh) factor | baseline to 24 weeks
  Change in Lung function Tests
Change in partial pressure of oxygen | baseline to 12 weeks
  Change in capillary or arterial blood gas analysis
Change in partial pressure of oxygen | baseline to 24 weeks
  Change in capillary or arterial blood gas analysis
Change in partial pressure of carbon dioxide | baseline to 12 weeks
  Change in capillary or arterial blood gas analysis
Change in partial pressure of carbon dioxide | baseline to 24 weeks
  Change in capillary or arterial blood gas analysis
Change in SaO2 | baseline to 12 weeks
  Change in capillary or arterial blood gas analysis
Change in SaO2 | baseline to 24 weeks
  Change in capillary or arterial blood gas analysis
Change in pH | baseline to 24 weeks
  Change in capillary or arterial blood gas analysis
Change in pH | baseline to 12 weeks
  Change in capillary or arterial blood gas analysis
Change in Blood pressure | baseline to 12 weeks
  Change in Cardiopulmonary exercise testing
Change in Blood pressure | baseline to 24 weeks
  Change in Cardiopulmonary exercise testing
Change in heart rate | baseline to 12 weeks
  Change in Cardiopulmonary exercise testing
Change in heart rate | baseline to 24 weeks
  Change in Cardiopulmonary exercise testing
Change in workload | baseline to 12 weeks
  Change in Cardiopulmonary exercise testing
Change in workload | baseline to 24 weeks
  Change in Cardiopulmonary exercise testing
Change in oxygen consumption as total and per kg body weight | baseline to 12 weeks
  Change in Cardiopulmonary exercise testing
Change in oxygen consumption as total and per kg body weight | baseline to 24 weeks
  Change in Cardiopulmonary exercise testing
Change in exhaled carbon dioxide (VCO2) | baseline to 12 weeks
  Change in Cardiopulmonary exercise testing
Change in exhaled carbon dioxide (VCO2) | baseline to 24 weeks
  Change in Cardiopulmonary exercise testing
Change in oxygen saturation | baseline to 12 weeks
  Change in Cardiopulmonary exercise testing
Change in oxygen saturation | baseline to 24 weeks
  Change in Cardiopulmonary exercise testing
Change in oxygen pulse | baseline to 12 weeks
  Change in Cardiopulmonary exercise testing
Change in oxygen pulse | baseline to 24 weeks
  Change in Cardiopulmonary exercise testing
Change in minute ventilation | baseline to 12 weeks
  Change in Cardiopulmonary exercise testing
Change in minute ventilation | baseline to 24 weeks
  Change in Cardiopulmonary exercise testing
Change in respiratory equivalents for oxygen | baseline to 12 weeks
  Change in Cardiopulmonary exercise testing
Change in respiratory equivalents for oxygen | baseline to 24 weeks
  Change in Cardiopulmonary exercise testing
Change in respiratory equivalents for carbon dioxide | baseline to 12 weeks
  Change in Cardiopulmonary exercise testing
Change in respiratory equivalents for carbon dioxide | baseline to 24 weeks
  Change in Cardiopulmonary exercise testing
Change in respiratory reserve | baseline to 12 weeks
  Change in Cardiopulmonary exercise testing
Change in respiratory reserve | baseline to 24 weeks
  Change in Cardiopulmonary exercise testing
WHO FC | baseline to 12 weeks
  Change in WHO functional class
WHO FC | baseline to 24 weeks
  Change in WHO functional class
SF-36 | baseline to 24 weeks
  Change in Quality of life parameters by questionnaire SF-36
NT-proBNP | baseline to 12 weeks
  Change in laboratory parameters
NT-proBNP | baseline to 24 weeks
  Change in laboratory parameters
haemoglobin changes | baseline to 12 weeks
  Change in laboratory parameters
haemoglobin changes | baseline to 24 weeks
  Change in laboratory parameters
haematocrit changes | baseline to 12 weeks
  Change in laboratory parameters
haematocrit changes | baseline to 24 weeks
  Change in laboratory parameters
AST changes | baseline to 12 weeks
  Change in liver enzymes
AST changes | baseline to 24 weeks
  Change in liver enzymes
ALT changes | baseline to 12 weeks
  Change in liver enzymes
ALT changes | baseline to 24 weeks
  Change in liver enzymes
Bilirubin changes | baseline to 12 weeks
  Change in liver enzymes
Bilirubin changes | baseline to 24 weeks
  Change in liver enzymes
CRP changes | baseline to 12 weeks
  Change in laboratory parameters
CRP changes | baseline to 24 weeks
  Change in laboratory parameters
sodium changes | baseline to 12 weeks
  Change in laboratory parameters
sodium changes | baseline to 24 weeks
  Change in laboratory parameters
Urea changes | baseline to 12 weeks
  Change in renal parameters
Urea changes | baseline to 24 weeks
  Change in renal parameters
creatinine changes | baseline to 12 weeks
  Change in renal parameters
creatinine clearance changes | baseline to 12 weeks
  Change in renal parameters
creatinine changes | baseline to 24 weeks
  Change in renal parameters
creatinine clearance changes | baseline to 24 weeks
  Change in renal parameters

CONTACTS AND LOCATIONS:
Overall Officials: Ekkehard HD Grünig, MD, Principal Investigator — Thoraxklinik at the University of Heidelberg
Locations (1):
- Centre for Pulmonary Hypertension at the Thoraxklinik Heidelberg, Heidelberg University Hospital, Heidelberg, Germany

REFERENCES:
- [Background] Raymond RJ, Hinderliter AL, Willis PW, Ralph D, Caldwell EJ, Williams W, Ettinger NA, Hill NS, Summer WR, de Boisblanc B, Schwartz T, Koch G, Clayton LM, Jobsis MM, Crow JW, Long W. Echocardiographic predictors of adverse outcomes in primary pulmonary hypertension. J Am Coll Cardiol. 2002 Apr 3;39(7):1214-9. doi: 10.1016/s0735-1097(02)01744-8. PMID 11923049
- [Background] Bossone E, D'Andrea A, D'Alto M, Citro R, Argiento P, Ferrara F, Cittadini A, Rubenfire M, Naeije R. Echocardiography in pulmonary arterial hypertension: from diagnosis to prognosis. J Am Soc Echocardiogr. 2013 Jan;26(1):1-14. doi: 10.1016/j.echo.2012.10.009. Epub 2012 Nov 8. PMID 23140849
- [Background] Austin C, Alassas K, Burger C, Safford R, Pagan R, Duello K, Kumar P, Zeiger T, Shapiro B. Echocardiographic assessment of estimated right atrial pressure and size predicts mortality in pulmonary arterial hypertension. Chest. 2015 Jan;147(1):198-208. doi: 10.1378/chest.13-3035. PMID 25211049
- [Background] Marra AM, Egenlauf B, Ehlken N, Fischer C, Eichstaedt C, Nagel C, Bossone E, Cittadini A, Halank M, Gall H, Olsson KM, Lange TJ, Grunig E. Change of right heart size and function by long-term therapy with riociguat in patients with pulmonary arterial hypertension and chronic thromboembolic pulmonary hypertension. Int J Cardiol. 2015 Sep 15;195:19-26. doi: 10.1016/j.ijcard.2015.05.105. Epub 2015 May 19. PMID 26011408
- [Background] Marra AM, Halank M, Benjamin N, Bossone E, Cittadini A, Eichstaedt CA, Egenlauf B, Harutyunova S, Fischer C, Gall H, Ghofrani HA, Hoeper MM, Lange TJ, Olsson KM, Klose H, Grunig E. Right ventricular size and function under riociguat in pulmonary arterial hypertension and chronic thromboembolic pulmonary hypertension (the RIVER study). Respir Res. 2018 Dec 19;19(1):258. doi: 10.1186/s12931-018-0957-y. PMID 30567595